CLINICAL TRIAL: NCT03212339
Title: Project BELONG: Breaking the Cycle of Intergenerational Family Violence and Trauma: Innovating, Expanding and Sustaining Treatment for Caregivers and Very Young Children
Brief Title: Project BELONG: Breaking the Cycle of Intergenerational Family Violence and Trauma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was halted due to challenges with recruitment and enrollment.
Sponsor: Boston Medical Center (Other)
Collaborators: The New School for Social Research (Other); Children's Bureau - Administration for Children and Families (Other)
Responsible Party: Principal Investigator, Neena McConnico, Program Director, Child Witness to Violence Project, Boston Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-35778; 90EV0450-01-00 (Other Grant/Funding Number: Family and Youth Services Bureau, DHHS)
Record Dates: First submitted 2017-05-30; First posted 2017-07-11 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Mother-child Relations; Parenting; Parent Child Abuse; Family Conflict; Parental Stress; Family Relations; Childhood Disorder of Social Functioning, Unspecified
Keywords: parent-child interactions; mental health care; child health services; parenting confidence; adverse childhood events; dyadic care model
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mothers with children <3 years of age (Experimental): Dyads of mothers with children up to 3 years of age will be attending modified Group Attachment Based Intervention (mGABI) sessions at the SPARK Center that will include a small group of other mother-child pairs and approximately two therapists. Dyads will be offered the 10 session therapeutic intervention.
  Interventions: Other: Therapeutic intervention
- Mothers with children 3-5 years of age (Experimental): Dyads of mothers with children between the ages of 3 and 5 years will be attending Brief Dyadic Intervention (BDI) sessions at Child Witness to Violence and/or the SPARK Center with their child and an individual therapist. Dyads will be offered the 10 session therapeutic intervention.
  Interventions: Other: Therapeutic intervention

INTERVENTIONS:
Other: Therapeutic intervention — Therapeutic interventions will be delivered in ten 2-hour sessions over 12-15 weeks, which includes 2 research data collection sessions at the beginning of the study (pre-intervention) and at the end of the study (post-intervention). During the pre-intervention data collection session, participants will be asked to provide demographic information and complete interviews about their past experiences and current experiences as a parent, and their child's current functioning. Parents will also be video recorded interacting with their child for 10 minutes. During the post-intervention data collection session, participants will be asked to complete a similar set of interviews and will also be video recorded interacting with their child for 10 minutes.

SUMMARY:
This study will examine the efficacy of a dyadic therapy intervention for mothers who have histories of adverse events (e.g., history of family violence, partner violence, family conflict, and/or childhood trauma, including abuse/neglect) and their very young children (ages 0-5 years), with the goal of demonstrating how an evidence supported, community-based and/or hospital-based therapeutic intervention may help reduce exposure to trauma and incidents of child maltreatment, improve parental stress and mental health, and secure parent-child attachment.

The three main objectives associated with Project BELONG are: 1) to determine the effectiveness of a dyadic care model in improving parent/child interaction, parenting confidence and competence, reducing parenting stress and social isolation, and improving access to concrete supports; 2) to address maltreatment risk in children by enhancing social-emotional functioning and developmental progress; and 3) to train new and future mental health professionals in dyadic mental health services and disseminate the model and findings through health professional schools and publications.

DETAILED DESCRIPTION:
A maximum of ninety (N=90) women and children will be screened and recruited from three clinical care programs at Boston Medical Center (BMC): 1) the SPARK Center, 2) Child Witness to Violence, and 3) Project RESPECT, to participate in therapeutic programming delivered by trained psychologists, social workers and therapists at the SPARK Center in Mattapan, MA or at Child Witness to Violence at BMC in Boston, MA. Mothers with children through the age of 3 years will be attending modified Group Attachment Based Intervention (mGABI) sessions at the SPARK Center that will include a small group of other mother-child pairs and approximately two therapists. Mothers with children between the ages of 3 and 5 years will be attending Brief Dyadic Intervention (BDI) sessions at Child Witness to Violence and/or the SPARK Center with their child and an individual therapist. The therapeutic interventions will be similar between the two groups and will be delivered in 10 sessions over the course of approximately 12-15 weeks. Each session will be approximately 2 hours long and will be scheduled to accommodate the participants' schedules. Participants will be asked to attend 1 session per week and to participate in two research data collection sessions that are part of the 10-session commitment. The first session will occur at the beginning of the study (pre-intervention) and the second session will occur at the end of the study (post-intervention). During the first data collection session, participants will be asked to provide demographic information and complete interviews about past experiences and current experiences as a parent, and their child's current functioning. Parents will also be video recorded interacting with their child for 10 minutes. During the second data collection session, participants will be asked to complete a similar set of interviews and they will be video recorded again interacting with their child for 10 minutes.

Project BELONG will address the impact of trauma and dyadic therapy on the mother and child as it affects parenting, child development, and child behavior. Changes in parents' ability to interact with their child in nurturing and responsive ways (as measured by coding videotapes of pre- and post- mother-child interactions) will be investigated as well as improvements in maternal symptoms of stress, depression and feelings of self-efficacy (as measured by validated, evidence-based pre- and post- assessments). Child outcomes will be assessed via change from baseline in measures of child's psychosocial functioning and development.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* 18 years of age or older
* Has a child under the age of 5 years
* Must be parent or legal guardian of child
* Comfortable communicating in English
* Plan to stay in the greater Boston area for the next 6 months [post IRB-approval]
* Typically available between the hours of 8:00 AM and 5:00 PM at least one day during the week (Monday thru Friday)
* Must answer "yes" to having experienced hardships in their own life, which may have involved any of the following: threat of violence, family violence, partner violence, family conflict, and/or mistreatment in their own childhood.
* Must be able to provide informed consent

Exclusion Criteria:

* Child previously diagnosed with autism, severe global delay, blindness, deafness or paralysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Parent-child interaction | Change from baseline and 14 weeks
  Parent-child interactions will be assessed from the 10-minute video recordings of naturalistic interaction between parent and child using the Coding Interactive Behavior (CIB) global rating system. The CIB assesses parent, child and dyadic affective states and interactive styles to measure social behavior. It includes multiple scales (ranging from 34 to 52 depending on age) organized into several composites that index important aspects of any relationship, such as sensitivity, intrusiveness, engagement, reciprocity.

SECONDARY OUTCOMES:
Parental concern of child development | week 1
  Parental concern of child development will be assessed via the 10-item Parent's Evaluation of Developmental Status (PEDS). The PEDS is an evidence-based method for detecting and addressing developmental and behavioral problems in children aged from birth to eight years. All responses are based on the age of the child and scoring sorts children into high, moderate or low risk for an undiagnosed developmental disability and behavioral problems requiring referral for in-depth evaluation.
Parenting stress | Change from baseline and 14 weeks
  Parenting stress will be assessed via the 36-item Parenting Stress Index (PSI) Short Form. The PSI is a screening and triage measure for evaluating the parenting system and identifying issues in parental functioning that may lead to problems in the child's behavior. Designed for use with parents of children ranging in age from 1 month to 12 years, the PSI yields a total stress score from three scales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child, using a 5-point scale ranging from strongly agree [1] to strongly disagree [5]. Scores are calculated for each sub-scales and then added to yield the Total Stress score. Altogether, the higher the score, the greater the level of stress in parents.
Parenting satisfaction and efficacy | Change from baseline and 14 weeks
  Parenting satisfaction and efficacy will be assessed via the 17-item Parenting Sense of Competence Scale (PSOC). The PSOC was designed to measure parental competence on two dimensions: satisfaction and efficacy, using a 6-point scale ranging from strongly agree [1] to strongly disagree [6], with ten questions under Satisfaction and seven under Efficacy. Satisfaction section examines the parents' anxiety, motivation and frustration, while the Efficacy section looks at the parents' competence, capability levels, and problem-solving abilities in their parental role. Scores are calculated by adding all responses to yield the participants PSOC score. A higher score indicates a higher parenting sense of competency; there are no average scores or 'cut-off's' for this tool.
Parental distress and depression | Change from baseline and 14 weeks
  Parental psychological distress, interpersonal sensitivity, and depression will be assessed via the 53-item Brief Symptom Inventory (BSI). The BSI was designed to evaluate psychological distress in the past week using a 4-point scale ranging from not at all [0] to extreme [4]. It is composed of nine primary symptom dimensions (somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism) and includes three global indices of distress (Global Severity, Positive Symptom Distress, and Positive Symptom Total) to measure the overall distress level, intensity of symptoms, and number of self-reported symptoms. A clinically significant score can be reached in two ways: the GSI score is greater than or equal to a T score of 63, or any two subscales are greater than or equal to a T score of 63 when compared with the norms for the particular population in question.
Parental reflective functioning | Change from baseline and 14 weeks
  Parental mentalization and reflective functioning will be assessed via the 18-item Parental Reflective Functioning Questionnaire (PRFQ). The PRFQ was designed for parents of children 0-5 years to provide a brief, multidimensional assessment of parental reflective functioning and mentalization, which refers to the caregiver's capacity to reflect upon her own internal mental experiences as well as those of the child. Parental reflective functioning is assumed to play a key role in fostering the developing child's own capacity for mentalizing, which in turn is important for the development of emotion regulation, a sense of personal agency, and secure attachment relationships. Items were formulated positively (i.e., higher scores reflect higher levels of parental reflective functioning) and negatively (i.e, higher scores reflect lower levels of mentalization).
Parental perceptions of infant/child development | Change from baseline and 14 weeks
  Parental perceptions of their infant/child development will be assessed via 6 questions adapted from the Working Model of the Child Interview (WMCI). The WMCI is a semi-structured, open-ended interview designed to assess parent's perception of and relationship with their infant/child. The questions adapted from the WMCI include: 1) "What are three things you feel are unique and different about your child compared to (what you know of) children?" 2) "What are three things that pleases you the most about your relationship with your child/baby?" 3) "Think for a moment of your child as an adult. What five hopes and fears do you have about that time?" 4) Pick 5 words to describe your impression of your child's personality now. 5) At this point, who does your child remind you of? In what ways? 6) Pick 5 words to describe your relationship with your child now. There is no score or 'cut-off' for this tool.
Parental childhood experiences of abuse and neglect | week 1
  Parental childhood experiences of abuse and neglect will be assessed via the 26-item Clinical Adverse Childhood Experience Questionnaire. The Clinical ACEs was adapted from the original ACEs Questionnaire and includes ten categories of childhood adversity: exposure to psychological, physical and sexual abuse, emotional and physical neglect, household dysfunction including parental divorce or separation, untreated parental mental illness, parental alcohol or substance abuse, parental incarceration, and exposure to mother treated violently. Scores are calculated by adding all responses to yield the participants PSOC score. A higher score indicates a higher risk of health and social problems; there are no average scores or 'cut-off's' for this tool.
Child social and emotional skills and competencies | Change from baseline and 14 weeks
  Child social and emotional skills and competencies will be assessed via the age-appropriate Devereux Early Childhood Assessment (DECA). The DECA is a standardized, strength based assessment to assess protective factors and screening for potential risks in the social and emotional development of very young children. The DECA Infant (4 weeks up to 18 months) has 33 items and comprises of two protective factor scales: Initiative and Attachment/Relationships. The DECA Toddler (age 18 months to 36 months) has 36 items and comprises of three protective factor scales: Initiative, Attachment/Relationships, and Self-Regulation. The DECA for Preschoolers (ages 3 to 6 years) has 38 items and comprises of four protective factor scales: Total protective Factors, Initiative, Self-Regulation, and Attachment/Relationships. Scores correspond to the child's age and rater, and are calculated by adding all responses in each scale. Scores place children in three categories: typical, strength, and concern.
Interviewer-observed parent-child interaction | Change from baseline and 14 weeks
  In addition to the 10-minute video recordings of naturalistic interaction between parent and child, parent-child interaction will be assessed via the interviewer-observed 8-item Home Observation Measurement of the Environment (HOME). The HOME was designed to measure the quality and quantity of stimulation and support available to a child in the home environment. There is no score or 'cut-off' for this tool.
Material hardships | Change from baseline and 14 weeks
  Food insecurity will be assessed via two standardized questions developed by the US Dept of Agriculture Economic Research: Guide to Measuring Household Food Security. These include "within the past 6 months…": 1) "…we worried whether our food would run out before we got money to buy more" and 2) "…the food we bought just didn't last and we didn't have money to get more." Housing instability will be assessed in accordance with previously published measures, as no official US measure exists. These include: 1) "What kind of housing do you currently live in?" 2) "Are you temporarily living with other people even for a little while because of financial difficulties?" 3) "Can you continue to stay where you are for as long as you want?" 4) "When was the last time if ever that you considered yourself to be without a regular place to stay or homeless?" and 5) "During the past 6 months, was there a time when you were not able to pay the mortgage/rent on time because of financial difficulties?"

CONTACTS AND LOCATIONS:
Overall Officials: Neena McConnico, PhD, LMHC, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No